CLINICAL TRIAL: NCT02560753
Title: Phase 2a Feasibility Study of T3D-959 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Feasibility Study in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: T3D Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T3D959-201
Record Dates: First submitted 2015-07-28; First posted 2015-09-25 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- T3D-959 3mg (Experimental): Nine subjects will take 3mg by mouth once daily for two weeks, with or without food.
  Interventions: Drug: T3D-959
- T3D-959 10mg (Experimental): Nine subjects will take 10mg by mouth once daily for two weeks, with or without food.
  Interventions: Drug: T3D-959
- T3D-959 30mg (Experimental): Nine subjects will take 30mg by mouth once daily for two weeks, with or without food.
  Interventions: Drug: T3D-959
- T3D-959 90mg (Experimental): Nine subjects will take 90mg by mouth once daily for two weeks, with or without food.
  Interventions: Drug: T3D-959

INTERVENTIONS:
Drug: T3D-959 — The 3mg dosage is supplied as 1mg capsules (three capsules, taken once daily by mouth) The 10mg dosage is supplied as 5mg capsules (two capsules, taken once daily by mouth) The 30mg dosage is supplied as either 5mg or 15mg capsules (six 5mg capsules or two 15mg capsules taken once daily by mouth) The 90mg dosage is supplied as 15mg capsules (six capsules, taken once daily by mouth)

SUMMARY:
The study is a randomized, parallel, 4-dose design in subjects with mild-to-moderate Alzheimer's Disease. Subjects will be randomized to one of 4 doses of T3D-959. Subjects will be evaluated for changes from baseline in cerebral metabolic rate of glucose (FDG-PET imaging), functional connectivity of the hippocampus (BOLD-fMRI), and cognitive function (ADAS-Cog11 and DSST) as well as assessed for safety and tolerability to T3D-959.

An expanded access extension is planed to provide access to study medication to subjects who have completed the main study and requested continued use.

DETAILED DESCRIPTION:
T3D-959 is an orally-delivered, once-a-day administered, small molecule dual nuclear receptor agonist that has been shown in animal and Phase 1 studies in normal human subjects to be safe and well tolerated. The purpose of this clinical study in AD patients is to demonstrate mechanistic proof of concept that T3D-959, can produce desired changes in cerebral glucose metabolism and functional connectivity that may indicate potential for cognitive improvement. The therapeutic approach to be tested is based on two suppositions; (A) ameliorating multiple pathologies in the disease with a single therapy may provide a superior clinical benefit than therapeutic approaches which target a single pathology and (B) correcting insulin resistance in the brain, (highly correlated with AD and potential key driver of AD pathophysiology) and peripherally may be disease remedial.

The brain requires integral insulin signaling for metabolic homeostasis and neuronal plasticity. Insulin resistance disrupts energy balance and signaling networks needed for a broad range of functions. Impaired insulin signaling in neurons enhances apoptosis, promotes oxidative cell death induced by Abeta1-42, increases secretion of Abeta1-42, blocks removal of extracellular Abeta oligomers and increases plaque loads. A growing body of evidence suggests that brain insulin resistance promotes or possibly is the trigger of key pathologies in AD and is supported by observed changes in levels of insulin signaling molecules in AD forebrains and associated changes in memory. Pre-clinical studies in animals have demonstrated the insulin sensitizing activity of T3D-959 and ability to improve multiple pathologies of AD in a rat model of disease.

This non-placebo controlled trial will be conducted in one to three clinical centers. Thirty six (36) patients with mild-to-moderate Alzheimer's disease will be randomly assigned to once daily, orally administered treatment with 3mg, 10mg, 30mg or 90mg doses of T3D-959. Participants will be treated for two weeks and will undergo at baseline and at two weeks; FDG-PET scans to measure brain glucose metabolism, BOLD fMRI scans to measure functional connectivity of the hippocampus, venous blood draws for biomarker analysis and ApoE genotyping, and ADAS-Cog11 and DSST cognitive testing. For monitoring potential toxicities of the drug subjects will undergo physical examination, neurological examination, adverse event review, blood chemistries, and pharmacokinetic (PK) analyses for T3D-959 plasma levels.

BOLD fMRI definition of terms:

GoF (Goodness of Fit): The degree to which the spatial extent and magnitude of one subject's default mode network (DMN) regions matches the one of an elderly control group.

Hippo-PreC Link (Hippocampus - Precuneus Link): The resting-state BOLD signal correlation strength between hippocampus and precuneus regions of interest.

GlobEff_DMN: (Global Efficiency from DMN Regions): The global efficiency among 11 pre-defined default mode network regions.

GlobEff_AAL: (Global Efficiency from AAL Regions): The global efficiency among 90 pre-defined cerebral regions based on automated anatomical labeling.

ALFF_lPCC_PreC: Amplitude of Low Frequency Fluctuations (ALFF) from left posterior cingulate cortex (PCC) and precuneus (PreC).

ALFF_rPCC_PreC: ALFF from right PCC and precuneus. fALFF_lPCC_PreC: Ratio ALFF from left PCC and precuneus. fALFF_rPCC_PreC: Ratio ALFF from right PCC and precuneus. ReHo_lPCC_PreC: Regional Homogeneity in left PCC and PreC. ReHo_rPCC_PreC: Regional Homogeneity in right PCC and PreC. ALFF_lIPL: ALFF from left inferior parietal lobule (IPL). ALFF_rIPL: ALFF from right IPL. fALFF_lIPL: Ratio ALFF from left IPL. fALFF_rIPL : Ratio ALFF from right IPL. ReHo_lIPL: Regional Homogeneity in left IPL. ReHo_rIPL: Regional Homogeneity in right IPL.

Expanded Access Extension: This is an open label 10 visit extension for up to 5 subjects who have completed the T3D959-201 protocol and whose caregivers and physician requested their continued treatment in an expanded access protocol. All subjects enrolled in this study will be treated with a 15mg q.d. dose of T3D959 for six months, regardless of their assigned dose level from the main study. A continued risk/benefit assessment by the investigator will be conducted at each visit to determine the need for treatment continuation. Subjects will be assessed for safety and tolerability to T3D-959 and evaluated for changes from baseline cognitive function via ADAS-Cog11 and DSST testing and global change via CIBIC-plus testing.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for mild-to-moderate AD with Mini-Mental State Examination (MMSE) score of 14 through 26
* Clinical Dementia Rating = 0.5 to 2.0
* Modified Hachinski less than or equal to 4
* A clinical diagnosis of AD per NINCDS-ADRDA criteria
* Washout of psychoactive medication (other than anti-depressants): at least 4 weeks prior to baseline
* Stability of all permitted medications for 4-12 weeks prior to baseline
* Visual and auditory acuity adequate for neuropsychological testing
* Home monitoring available for supervision of medications

Exclusion Criteria:

* Unstable diabetes or insulin use
* Unable to participate in FDG-PET scanning
* Inability to undergo a clinical MRI of the brain
* Diagnosis of significant neurological/psychiatric disease other than AD
* History of moderate or severe congestive heart failure, NYHA class III or IV, within 12 months prior to baseline.
* Previous cardiovascular event within the past 6 months prior to baseline
* Subject is pregnant, or lactating.
* ALT and/or AST levels that are twice the upper limit of normal; bilirubin levels that exceed 2 mg/dL; serum creatinine >1.5 mg/dL in men or > 1.4 mg/dL in women.
* Current or history of severe or unstable disorder (medical or psychiatric) requiring treatment that may make the subject unlikely to complete the study.
* Current use of fluvoxamine.
* Current unstable use of warfarin.
* Current use (within 30 days of baseline, visit 2) of certain highly protein-bound medications
* Malignancy within the last 5 years (other than non-melanoma skin cancer, stable, non-progressive prostate cancer not requiring treatment or in situ cervical cancer).
* Known history of HIV, hepatitis B, or hepatitis C.
* Blood pressure greater than 160/100 mmHg.
* Known or suspected intolerance or hypersensitivity to the study drugs, closely related compounds, or any of their stated ingredients.
* History of alcohol, drug abuse or dependence (except nicotine dependence) within 2 years.
* Investigational amyloid lowering therapies use within two months prior to baseline
* Have participated in any other investigational study or received an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to baseline
* Any surgical or medical condition which may significantly alter the absorption of any drug substance
* Resides in hospital or moderate to high dependency continuous care facility.
* Non ambulatory, or wheelchair-bound
* History of swallowing difficulties.
* Evidence of clinically relevant pathology that in the investigator's opinion could interfere with the study results or put the subject's safety at risk.

Expanded Access Extension :

Subjects must continue to meet the main study inclusion/exclusion criteria to insure continued safety to continue on a 6 months study extension

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Didsbury, Ph.D., Study Chair — T3DTherapeutics, Inc.
Locations (3):
- United States (3):
  - Brain Matters Research, Delray Beach, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - New Hope Clinical Research, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tong M, Dominguez C, Didsbury J, de la Monte SM. Targeting Alzheimer's Disease Neuro-Metabolic Dysfunction with a Small Molecule Nuclear Receptor Agonist (T3D-959) Reverses Disease Pathologies. J Alzheimers Dis Parkinsonism. 2016 Jun;6(3):238. doi: 10.4172/2161-0460.1000238. Epub 2016 Jun 3. PMID 27525190
- [Derived] Tong M, Deochand C, Didsbury J, de la Monte SM. T3D-959: A Multi-Faceted Disease Remedial Drug Candidate for the Treatment of Alzheimer's Disease. J Alzheimers Dis. 2016;51(1):123-38. doi: 10.3233/JAD-151013. PMID 26836193

RESULTS

PARTICIPANT FLOW:
Groups:
- T3D-959 3mg: subjects took 3mg by mouth once daily for two weeks, with or without food.
  T3D-959: The 3mg dosage was supplied as 1mg capsules (three capsules, taken once daily by mouth)
- T3D-959 10mg: subjects took 10mg by mouth once daily for two weeks, with or without food.
  The 10mg dosage was supplied as 5mg capsules (two capsules, taken once daily by mouth)
- T3D-959 30mg: subjects took 30mg by mouth once daily for two weeks, with or without food.
  The 30mg dosage was supplied as either 5mg or 15mg capsules (six 5mg capsules or two 15mg capsules taken once daily by mouth)
- T3D-959 90mg: subjects took 90mg by mouth once daily for two weeks, with or without food.
  The 90mg dosage was supplied as 15mg capsules (six capsules, taken once daily by mouth)
Period: Overall Study
Arm/Group | T3D-959 3mg | T3D-959 10mg | T3D-959 30mg | T3D-959 90mg
Started | 9 | 9 | 10 | 8
Completed | 8 | 9 | 9 | 8
Not Completed | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T3D-959 3mg | T3D-959 10mg | T3D-959 30mg | T3D-959 90mg | Total
Number analyzed (Participants) | 9 | 9 | 10 | 8 | 36
Age, Customized [Count of Participants; unit: Participants]
  <=65 years | 2 | 2 | 3 | 1 | 8
  65-74 years | 2 | 4 | 2 | 2 | 10
  75-84 years | 3 | 3 | 1 | 5 | 12
  >84 years | 2 | 0 | 4 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 4 | 20
  Male | 4 | 4 | 4 | 4 | 16
ApoE4 genotype [Count of Participants; unit: Participants] — Population: This measure is assessed on study completers
  Participants
    number analyzed (Participants) | 8 | 9 | 9 | 8 | 34
    ApoE4 positive | 4 | 2 | 4 | 3 | 13
    ApoE4 negative | 4 | 7 | 5 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (End of Treatment - Baseline) for FDG-PET Imaging With Whole Brain and White Matter as Reference Region
Description: Changes in relative brain glucose metabolism (delta R CMRgl) were measured by FDG-PET. At each time point, a ratio of the PET reading in a pre-defined region of interest (sROI), known to be affected by AD, and in a reference region (RR) that is spared in AD, is determined. This ratio is defined as "sROI index" (spared region). A second RR, brain white matter (WM), was also used in this calculation: sROI index" (WM) value. delta sROI is defined as change in the sROI index values, over the treatment period. In this study we are looking for changes in delta sROI with increasing doses of T3D-959. Dose dependent changes in delta sROI (AD spared) are compared to those observed with the WM as the RR: delta sROI (WM). Dose related changes in delta sROI suggests T3D-959 is entering the brain and effecting glucose metabolism in a dose dependent fashion.
Time Frame: after 14 days of treatment
Population: Both + & - values for delta sROI represent "better outcomes" with regard to the demonstrating pharmacological activity of a PPAR delta, such as T3D-959, in the brain. It is unknown at this time, both from this presented data and from the literature, whether the pharmacological action of a PPAR delta agonist will translate to better outcomes in AD.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | T3D-959 3mg | T3D-959 10mg | T3D-959 30mg | T3D-959 90mg
Number analyzed (Participants) | 9 | 9 | 10 | 8
ratio
  delta sROI (AD spared) | 0.0015 (0.02057) | 0.0034 (0.01671) | -0.0204 (0.01952) | -0.0293 (0.01744)
  delta sROI (white matter) | 0.0016 (0.04008) | 0.0053 (0.02471) | -0.0200 (0.01979) | -0.0355 (0.02303)

2. Primary Outcome: The Effect of Treatment With T3D-959 on Changes in Resting State Blood Oxygen Level Dependent (BOLD) Signal in Functional Magnetic Resonance Imaging (fMRI) of the Brain Areas Associated With Cognitive Tasks.
Description: Changes in BOLD fMRI parameters such as GoF (see Study Description) over the course of two weeks of treatment, were obtained in this study. BOLD fMRI has been used in cross sectional and longitudinal studies of Alzheimer's subjects, for instance in the Alzheimer's Disease Neuroimaging Initiative studies. However, no studies monitoring Default Mode Networks measured parameters such as GoF, in the context of an effective AD therapeutic, as a result it is difficult to interpret the observed small changes listed in BOLD fMRI parameters obtained in this trial. Instead the changes in the listed BOLD fMRI parameters (EOT - BL) are reported without interpretation. These values represent changes in fMRI connectivity patterns over time and are unitless.
Time Frame: after 14 days of treatment
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | T3D-959 3mg | T3D-959 10mg | T3D-959 30mg | T3D-959 90mg
Number analyzed (Participants) | 8 | 9 | 9 | 8
unitless
  GoF (Goodness of Fit) | 0.0129 (0.08528) | -0.0120 (0.0646) | 0.0118 (0.03375) | 0.0076 (0.08755)
  Hippo-PreC Link (Hippocampus - Precuneus Link) | -0.1213 (0.17904) | 0.1320 (0.22964) | 0.1196 (0.23035) | -0.0349 (0.18496)
  GlobEff_DMN(Global Efficiency from DMN Regions) | 0.0033 (0.00734) | -0.0036 (0.00940) | -0.0004 (0.00926) | -0.0001 (0.00397)
  GlobEff_AAL(Global Efficiency from AAL Regions) | -0.0001 (0.00664) | -0.0006 (0.00972) | -0.0031 (0.01060) | -0.0005 (0.00517)
  ALFF_lPCC_PreC (Amplitude of Low Frequency Fluctua | -0.0578 (0.12314) | -0.0190 (0.11983) | -0.0505 (0.07463) | -0.0206 (0.10508)
  ALFF_rPCC_PreC (ALFF from right PCC and precuneus) | -0.0752 (0.09059) | -0.0127 (0.12127) | -0.0097 (0.08362) | -0.0325 (0.11092)
  fALFF_lPCC_PreC (Ratio ALFF from left PCC & prec | 0.0121 (0.03246) | 0.0068 (0.03510) | -0.0132 (0.03955) | -0.0167 (0.03284)
  fALFF_rPCC_PreC (Ratio ALFF from right PCC & pre | -0.0080 (0.04094) | 0.0084 (0.04325) | -0.0007 (0.03913) | -0.0118 (0.04236)
  ReHo_lPCC_PreC (Regional Homogeneity in left PCC a | -0.0665 (0.18502) | 0.0237 (0.14028) | -0.0369 (0.09702) | 0.0194 (0.20061)
  ReHo_rPCC_PreC (Regional Homogeneity in right PCC | -0.0390 (0.06406) | -0.0663 (0.22082) | -0.0895 (0.10541) | -0.0041 (0.15836)
  ALFF_lIPL (ALFF from left inferior parietal lobule | -0.0635 (0.09445) | 0.0104 (0.05763) | -0.0102 (0.12016) | -0.0401 (0.05657)
  ALFF_rIPL(ALFF from right IPL) | -0.0493 (0.11288) | -0.0276 (0.12720) | 0.0346 (0.09654) | -0.1089 (0.13935)
  fALFF_lIPL (Ratio ALFF from left IPL) | -0.0296 (0.03988) | 0.0164 (0.02269) | -0.0107 (0.06563) | -0.0350 (0.04570)
  fALFF_rIPL (Ratio ALFF from right IPL) | -0.0342 (0.03912) | 0.0061 (0.03286) | 0.0023 (0.02771) | -0.0395 (0.05327)
  ReHo_lIPL (Regional Homogeneity in left IPL) | -0.0694 (0.15420) | 0.0147 (0.14620) | -0.0249 (0.19178) | -0.0062 (0.06575)
  ReHo_rIPL (Regional Homogeneity in right IPL) | -0.0694 (0.15420) | 0.0147 (0.14620) | -0.0249 (0.19178) | -0.0062 (0.06575)

3. Secondary Outcome: Change From Baseline in the Score of the Digit Symbol Substitution Test
Description: The digit symbol substitution test assesses attention, psychomotor speed, complex scanning, visual tracking, and immediate memory. This test consists of 4 rows each with 25 small blank squares; above each square is a number between 1 and 9. At the top is a 'key,' which pairs each number (1 through 9) with an unfamiliar symbol. The participant has 90 seconds to work as quickly as possible (left to right across the rows) to fill in each blank square with the appropriate symbol based on the number above the square. Results are presented as total number correct; therefore, lower numbers indicate greater impairment. Scores on the DSST range from 0-93.
Time Frame: after 14 days of treatment
Population: 3 mg group:A subject Dc'd prior to the EOT & another subject became uncooperative at EOT and refused to take the DSST. Her results for EOT were missing. 30 mg: A subject DC'd prior to EOT, another subject was described as being very agitated at the EOT. The results presented omitted this subject's EOT data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T3D-959 3mg | T3D-959 10mg | T3D-959 30mg | T3D-959 90mg
Number analyzed (Participants) | 9 | 9 | 10 | 8
score on a scale
  Change from baseline at end of treatment (day 14): number analyzed (Participants) | 7 | 9 | 8 | 8
  Change from baseline at end of treatment (day 14) | 4.429 (9.1626) | 1.000 (5.500) | 0.750 (3.6154) | 1.125 (4.5493)
  Change from baseline at follow-up (day 21): number analyzed (Participants) | 8 | 9 | 9 | 8
  Change from baseline at follow-up (day 21) | 5.375 (8.5011) | 3.111 (5.0111) | 4.000 (5.6789) | 6.625 (11.4385)

4. Secondary Outcome: Change From Baseline in the Total Score of the 11-item Alzheimer's Disease Assessment Scale - Cognitive Subscale
Description: The 11-item Alzheimer's Disease Assessment Scale (ADAS-Cog 11) is a psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis. The score can range between 0 and 70. A higher score indicates more cognitive impairment. A positive change in the score indicates cognitive worsening. The minimum severity score is 0 and the maximum severity score is 70.
Time Frame: after 14 days of treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T3D-959 3mg | T3D-959 10mg | T3D-959 30mg | T3D-959 90mg
Number analyzed (Participants) | 9 | 9 | 10 | 8
score on a scale
  Change from baseline at end of treatment (day 14): number analyzed (Participants) | 8 | 9 | 8 | 8
  Change from baseline at end of treatment (day 14) | -2.367 (4.0417) | -0.552 (3.1467) | -2.709 (3.9801) | 1.970 (5.2191)
  Change from baseline at follow-up (day 21): number analyzed (Participants) | 8 | 9 | 9 | 8
  Change from baseline at follow-up (day 21) | -3.409 (3.5168) | -0.624 (3.8134) | -4.119 (3.8163) | 2.795 (4.1567)

5. Other Pre Specified Outcome: Safety and Tolerability of Treatment With T3D-959 Over a 2-week Period in Subjects With Mild-to-moderate AD. New
Description: Number of participants with treatment related adverse events (AEs) as assessed by analysis of adverse events, including symptoms, and abnormal findings on physical and neurological examinations, and standard labs.
Time Frame: after 14 days of treatment
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | T3D-959 3mg | T3D-959 10mg | T3D-959 30mg | T3D-959 90mg
Number analyzed (Participants) | 9 | 9 | 10 | 8
participants
  Subjects with at Least One Serious Adverse Events | 0 | 0 | 0 | 0
  Subjects with at Least One Drug-related AE | 0 | 0 | 1 | 0
  Subjects with at Least One mild AE | 2 | 0 | 1 | 0
  Subjects with at Least One moderate AE | 1 | 0 | 2 | 0
  Subjects with at Least One serious AE | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: pre treatment, during the two weeks of treatment and on follow-up one week after treatment
Arm/Group | T3D-959 3mg | T3D-959 10mg | T3D-959 30mg | T3D-959 90mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 1/9 | 0/9 | 1/10 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T3D-959 3mg (N=9) | T3D-959 10mg (N=9) | T3D-959 30mg (N=10) | T3D-959 90mg (N=8)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No